CLINICAL TRIAL: NCT06757023
Title: A Clinical Follow-up Study on the Efficacy of Thumbtack Needle for Postoperative Sleep and Recovery Treatment
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Principal Investigator, Yang Bin, Principal Investigator, Fujian Medical University
Other Study IDs: FirstAHXiamenU-YB-3
Record Dates: First submitted 2024-12-18; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Postoperative Complications; Postoperative Pain; Acupuncture
MeSH Terms: conditions — Postoperative Complications; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing breast cancer surgery with general anesthesia in the hospital

SUMMARY:
To understand the impact of thumb-tack needle therapy on postoperative sleep and recovery in patients who have undergone general anesthesia, and to explore the clinical significance of thumb-tack needle therapy in improving postoperative sleep quality, preventing postoperative sleep disorders, and promoting postoperative recovery

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing breast cancer surgery with general anesthesia in the hospital;
2. American Society of Anesthesiologists (ASA) classification I-II;
3. Women aged 18-55 years;
4. No history of chronic insomnia;
5. Individuals who have not taken sedative-hypnotic drugs within the past month.

Exclusion Criteria:

1. Those who do not meet the aforementioned inclusion criteria;
2. A history of severe heart, brain, lung, or kidney diseases (such as acute coronary syndrome (ACS), severe heart failure classified as NYHA Class III or IV, severe arrhythmias, severe valvular disease; acute aortic disease, and severe peripheral vascular disease, etc.), or poor physical condition (including reduced exercise tolerance, multi-organ dysfunction, malnutrition, etc.);
3. A history of sleep disorders and psychiatric history;
4. Inability to receive thumb-tack needle treatment.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients undergoing breast cancer surgery with general anesthesia in the hospital
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2026-10-13 (Estimated); Study Completion 2026-11-13 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh sleep quality index(PSQI) | 1 day or 2 days before anesthesia exposure and 1, 3, and 7 days after anesthesia exposure.
  Total scores range from 0 to 21, with higher scores indicating worse sleep quality.

SECONDARY OUTCOMES:
Later Recovery evaluated by QoR-40 questionnaire | QoR-40 score on the third day after surgery
  The maximum total score is 200, with higher scores indicating better recovery quality

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No